CLINICAL TRIAL: NCT00070187
Title: A Phase II/III Study of Immunomodulation After High Dose Myeloablative Therapy With Autologous Stem Cell Rescue for Refractory/Relapsed Hodgkin Disease
Brief Title: Immunotherapy Using Cyclosporine, Interferon Gamma, and Interleukin-2 After High-Dose Myeloablative Chemotherapy With Autologous Stem Cell Transplantation in Treating Patients With Refractory or Relapsed Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHOD0121; CDR0000330135 (Other: Clinical Trials.gov); COG-AHOD0121 (Other: Children's Oncology Group)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Recurrence | interventions — aldesleukin; Interleukin-2; Filgrastim; Granulocyte Colony-Stimulating Factor; Interferon-gamma; interferon gamma-1b; interferon gamma, Cys(-3), Tyr(-2), Cys(-1)-; Carmustine; Cyclosporine; Cyclosporins; Cytarabine; Etoposide; etoposide phosphate; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperfractionated Involved-Field Radiotion-immunotherapy (Experimental): Completed prior salvage induction therapy and have not received full tissue tolerance from prior radiotherapy may receive hyperfractionated involved-field radiotherapy twice daily for 7 days.
  HIGH-DOSE PREPARATIVE REGIMEN: Beginning within 7 days after radiotherapy, carmustine IV over 3 hours on day -6; etoposide IV over 1 hour and cytarabine IV over 1 hour on days -5 to -2; and melphalan IV over 30 minutes on day -1.
  ASCT: Autologous bone marrow or peripheral blood stem cell transplantation on day 0. Filgrastim (oral or IV) beginning on day 1 and continuing until blood counts recover.
  IMMUNOTHERAPY: Cyclosporine IV twice daily beginning on day 0 and continuing until the completion of the course of recombinant interferon gamma and interleukin-2. When sufficiently recovered, Aldesleukin once daily for 18 days.
  Interventions: Biological: aldesleukin; Biological: filgrastim; Biological: recombinant interferon gamma; Drug: carmustine; Drug: cyclosporine; Drug: cytarabine; Drug: etoposide; Drug: melphalan; Procedure: autologous bone marrow transplantation; Procedure: bone marrow ablation with stem cell support; Procedure: peripheral blood stem cell transplantation
- Hyperfractionated Involved-Field Radiotion-no immunotherapy (Experimental): Completed prior salvage induction therapy and have not received full tissue tolerance from prior radiotherapy may receive hyperfractionated involved-field radiotherapy twice daily for 7 days.
  HIGH-DOSE PREPARATIVE REGIMEN: Beginning within 7 days after radiotherapy, carmustine IV over 3 hours on day -6; etoposide IV over 1 hour and cytarabine IV over 1 hour on days -5 to -2; and melphalan IV over 30 minutes on day -1.
  ASCT: Autologous bone marrow or peripheral blood stem cell transplantation on day 0. Filgrastim (oral or IV) beginning on day 1 and continuing until blood counts recover.
  Interventions: Biological: filgrastim; Drug: carmustine; Drug: cyclosporine; Drug: cytarabine; Drug: etoposide; Drug: melphalan; Procedure: autologous bone marrow transplantation; Procedure: bone marrow ablation with stem cell support; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: aldesleukin — Given IV
  Other Names: Proleukin; IL-2; recombinant human Interleukin 2; NSC # 373364
  Arms: Hyperfractionated Involved-Field Radiotion-immunotherapy
Biological: filgrastim — Given IV
  Other Names: GRANULOCYTE COLONY-STIMULATING FACTOR; r-metHuG-CSF; G-CSF; Neupogen; NSC #614629
Biological: recombinant interferon gamma — Given IV
  Other Names: INTERFERON GAMMA-1b; Actimmune; gamma interferon; immune interferon; lymphocyte interferon; rIFN-gamma; T-interferon; NSC #600662
  Arms: Hyperfractionated Involved-Field Radiotion-immunotherapy
Drug: carmustine — Given IV
  Other Names: BCNU; BiCNU; bischloronitrosourea; NSC #40996
Drug: cyclosporine — Given IV
  Other Names: cycloporine; Sandimmune; Neoral; Gengraf; NSC #290193
Drug: cytarabine — Given IV
  Other Names: cytosine arabinoside; AraC; Cytosar; NSC #063878
Drug: etoposide — Given IV
  Other Names: VP-16; VePesid; Etopophos; NSC #141540
Drug: melphalan — Given IV
  Other Names: L-PHENYLANINE mustard; L-PAM; L-sarcolysin; Alkeran; NSC #008806
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with autologous stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Giving immunotherapy using cyclosporine, interferon gamma, and interleukin-2 after stem cell transplantation may help the transplanted cells make an immune response and kill any remaining cancer cells. It is not yet known whether high-dose chemotherapy followed by autologous stem cell transplantation is more effective with or without immunotherapy.

PURPOSE: This randomized phase II/III trial is studying how well high-dose chemotherapy followed by autologous stem cell transplantation, cyclosporine, interferon gamma, and interleukin-2 works and compares it to high-dose chemotherapy followed by autologous stem cell transplantation only in treating patients with refractory or relapsed Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Phase II

  * Determine the feasibility and toxicity of immunotherapy comprising cyclosporine, interferon gamma, and interleukin-2 after high-dose myeloablative chemotherapy with autologous stem cell transplantation (ASCT) in patients with refractory or relapsed Hodgkin's lymphoma.

    * Phase II part of the study was completed and should have proceeded to Phase III; however long delay occurred due to some proposed protocol changes to Phase III , so long that the study got permanently closed ***********
* Phase III

  * Compare the event-free and overall survival of patients treated with vs without this immunotherapy regimen.

Secondary

* Determine the event-free and overall survival rates, toxic effects, and response rates to reinduction chemotherapy followed by hyperfractionated involved-field radiotherapy, high-dose chemotherapy comprising carmustine, etoposide, cytarabine, and melphalan, and ASCT in these patients.
* Correlate tumor biologic characteristics with response in patients treated with these regimens.
* Determine the effectiveness of this immunotherapy regimen in producing autologous graft-vs-host disease (GVHD) and auto-reactive cytotoxic T-lymphocyte activity in these patients.
* Correlate greater levels of autologous GVHD and in vitro cytolytic activity with improved event-free and overall survival in patients treated with these regimens.
* Determine whether treatment with immunotherapy can overcome the negative prognostic significance of p53 mutation and high serum levels of interleukin-10 and interleukin-2 receptor in these patients.
* Determine the genotoxicity of retrieval therapy and the incidence of hypermutability by longitudinal genotoxic biomonitoring in these patients.
* Correlate HLA class II invariant peptide (CLIP) expression in tumor cells with improved event-free and overall survival in patients treated with immunotherapy regimen.

OUTLINE: This is a nonrandomized, multicenter phase II study followed by a randomized, multicenter phase III study. Patients are stratified according to study phase (II vs III).

Patients receive 2 courses of salvage induction therapy on COG-AHOD00P1 or equivalent. Within 2-5 weeks after completion of salvage induction therapy, patients receive protocol therapy.

* Phase II: All patients receive the following treatment:

  * Hyperfractionated involved-field radiotherapy: Patients who have completed prior salvage induction therapy and have not received full tissue tolerance from prior radiotherapy may receive hyperfractionated involved-field radiotherapy twice daily for 7 days.
  * High-dose preparative regimen: Beginning within 7 days after radiotherapy, patients receive carmustine IV over 3 hours on day -6; etoposide IV over 1 hour and cytarabine IV over 1 hour on days -5 to -2; and melphalan IV over 30 minutes on day -1.
  * Autologous stem cell transplantation: Patients undergo autologous bone marrow or peripheral blood stem cell transplantation on day 0. Patients then receive filgrastim (G-CSF) subcutaneously (SC) or IV beginning on day 1 and continuing until blood counts recover.
  * Immunotherapy: Patients receive cyclosporine IV twice daily beginning on day 0 and continuing until the completion of the course of interferon gamma and interleukin-2. When sufficiently recovered, patients also receive interferon gamma SC every other day for 10 doses. Beginning 2 days after the start of interferon gamma, patients also receive interleukin-2 SC once daily for 18 days.
* Phase III: Patients who respond to prior salvage induction therapy are randomized to 1 of 2 treatment arms. Patients who have progressive disease after 2 courses of prior salvage induction therapy are assigned to arm I.

  * Arm I: Patients receive treatment as in phase II.
  * Arm II: Patients receive treatment as in phase II without immunotherapy. In both phases, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 year.

PROJECTED ACCRUAL: A total of 156 patients (25 for phase II and 131 for phase III) will be accrued for this study within 5.4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Hodgkin's lymphoma

  * Histologically confirmed at original diagnosis AND at relapse or disease progression
  * Relapsed or refractory to conventional therapy
* No recurrence without B symptoms or bulky disease at least 1 year after completion of minimal systemic therapy defined by either of the following:

  * Stage IA/IIA with nodal disease previously treated with radiotherapy only
  * Stage IA/IIA with nodal disease previously treated with less than 3 courses of standard dose chemotherapy
* Concurrently enrolled on the COG-AHOD00P1 salvage chemotherapy study OR received other appropriate salvage therapy (e.g., ifosfamide and vinorelbine)

PATIENT CHARACTERISTICS:

Age

* Under 30

Performance status

* ECOG 0-2 (for adults)
* Lansky 50-100% (for children)

Life expectancy

* At least 2 months

Hematopoietic

* Absolute neutrophil count at least 500/mm^3

Hepatic

* Bilirubin no greater than 1.5 times normal
* SGPT less than 2.5 times normal

Renal

* Creatinine no greater than 1.5 times normal OR
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min/1.73 m^2

Cardiovascular

* Shortening fraction at least 27% by echocardiogram OR
* Ejection fraction at least 50% by MUGA

Pulmonary

* No evidence of dyspnea at rest
* No exercise intolerance
* DLCO at least 50% (patients 8 years of age and over)

Other

* Not pregnant or nursing
* Negative pregnancy test
* No concurrent serious illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Recovered from prior immunotherapy
* At least 1 week since prior antineoplastic biologic agents
* More than 1 week since prior growth factors
* No prior stem cell transplantation
* No other concurrent immunomodulating agents

Chemotherapy

* See Disease Characteristics
* More than 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No other concurrent anticancer chemotherapy

Endocrine therapy

* No concurrent steroids, including dexamethasone as an antiemetic

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy

Surgery

* Not specified

Other

* No concurrent participation in another COG therapeutic study

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2003-11; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Incidence of death, excluding death due to disease, during the period of time from day 0 (transplant) through day 100 post transplant | Day 0 (transplant) through Day 100 (Post transplant)
  Death, excluding death due to disease, during the period of time from Day 0 (transplant) through Day 100 post transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Allen R. Chen, MD, PhD, MHS, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Sharon L. Gardner, MD, Study Chair — NYU Langone Health
Locations (63):
- United States (60):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital and Research Center - Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Children's Hospital of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - Hopital Sainte Justine, Montreal, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Chen AR, Hutchison R, Hess A, et al.: Clinical outcomes of patients with recurrent/refractory Hodgkin disease receiving cyclosporine, interferon-, and interleukin-2 immunotherapy to induce auto-reactivity after autologous stem cell transplantation with BEAM: a COG study. [Abstract] Blood 110 (11): A-1896, 2007.